CLINICAL TRIAL: NCT05293392
Title: Improving Pediatric COVID-19 Vaccine Awareness, Access, and Accountability in Underrepresented Communities
Brief Title: Improving COVID-19 Vaccine Uptake Among Black and Latino Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Health System (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); University of Delaware (Other); ChristianaCare (Other)
Responsible Party: Principal Investigator, Thao-Ly Phan, Associate Professor of Pediatrics; Research Scientist, Nemours Children's Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: U54GM104941-09S1 (NIH); U54GM104941-09S1 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-03-24 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: Healthcare disparities; Vaccine hesitancy
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally-Tailored COVID-19 Vaccine Uptake Intervention (Experimental)
  Interventions: Behavioral: Culturally-Tailored COVID-19 Vaccine Uptake Intervention
- Standard Care (Active Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Culturally-Tailored COVID-19 Vaccine Uptake Intervention — This is a multi-component intervention to increase COVID-19 vaccine uptake among youth that was co-created with community partners and refined with qualitative feedback from Black and Latino youth and parents. The intervention consists of culturally-tailored educational materials to increase awareness about the COVID-19 vaccine, culturally-sensitive communication strategies employed by pediatric primary care providers and community health workers, and strategies to facilitate and standardize access to the COVID-19 vaccine in the primary care clinic.
  Arms: Culturally-Tailored COVID-19 Vaccine Uptake Intervention
Behavioral: Standard Care — Standard care includes routine offer of the COVID-19 vaccine and counseling about the COVID-19 vaccine by pediatric primary care providers.
  Arms: Standard Care

SUMMARY:
Black and Latino youth may be less likely to get the COVID-19 vaccine than White youth. In this study we will work with community members to come up with ways to help Black and Latino families learn more about the COVID-19 vaccine and get the COVID-19 vaccine. We will test these ideas out in pediatric primary care clinics. This study will help us make sure that all youth have an equal chance of getting the COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Youth 0-21 years of age and their caregiver
* Receiving care at one of four Nemours primary care practices selected for this study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5792 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thao-Ly T Phan-Vo, MD, MPH, Principal Investigator — Nemours Children's Health
Locations (1):
- Nemours Children's Hospital, Delaware, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four primary care clinics were recruited to participate in the pilot cluster randomized clinical trial. Primary care clinics were randomized 1:1 to receive the intervention or not, with stratification by geographic region (Northern and Southern Delaware). Because of the cluster randomized nature of the trial and collection of data routinely collected in the electronic health record, a waiver of consent was approved.
Pre-assignment Details: Patients were counted as participants if they were eligible for but had not received the COVID-19 vaccine at the time of a visit to one of the participating clinics. Because individual patients were counted at the time of their clinic visit and the intervention was implemented in phases, participation differed from phase to phase. While the intervention was delivered to both patient (child) and their parent, only data about the patient (child) was collected from the electronic health record.
Units Other Than Participants: Primary care clinic
Period: Phase 1: Community-Tailored Handouts
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
Started | 268; 2 Primary care clinic | 406; 2 Primary care clinic
Completed | 268; 2 Primary care clinic | 406; 2 Primary care clinic
Not Completed | 0; 0 Primary care clinic | 0; 0 Primary care clinic
Period: Phase 2: Videos Featuring Local Families
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
Started | 281; 2 Primary care clinic | 476; 2 Primary care clinic
Completed | 281; 2 Primary care clinic | 476; 2 Primary care clinic
Not Completed | 0; 0 Primary care clinic | 0; 0 Primary care clinic
Period: Phase 3: Family-Centered Communication
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
Started | 442; 2 Primary care clinic | 628; 2 Primary care clinic
Completed | 442; 2 Primary care clinic | 628; 2 Primary care clinic
Not Completed | 0; 0 Primary care clinic | 0; 0 Primary care clinic
Period: Phase 4:Community Health Worker Outreach
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
Started | 1230; 2 Primary care clinic | 2019; 2 Primary care clinic
Completed | 1230; 2 Primary care clinic | 2019; 2 Primary care clinic
Not Completed | 0; 0 Primary care clinic | 0; 0 Primary care clinic

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care | Total
Number analyzed (Participants) | 2221 | 3529 | 5750
Age, Customized [Number; unit: participants]
  5-11 | 1268 | 1985 | 3253
  12-17 | 953 | 1544 | 2497
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1049 | 1736 | 2785
  Male | 1171 | 1793 | 2964
  Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 480 | 511 | 991
  Non-Hispanic Black | 627 | 1177 | 1804
  Non-Hispanic White | 923 | 1481 | 2404
  Non-Hispanic Other | 191 | 360 | 551
Region of Enrollment [Number; unit: participants]
  United States | 2221 | 3529 | 5750
COVID-19 vaccination rate in participating clinics in the month prior to trial [Number; unit: Percent of participants vaccinated] — Because this was a cluster randomized controlled trial, we analyzed each participating clinic's COVID-19 vaccination rate in the month prior to the start of the clinical trial to establish a baseline COVID-19 vaccination rate for the groups. In particular, we report the percent of participants vaccinated against COVID-19 at each clinic. Population: The number of participants represents the number of patients who had a visit to one of the participating primary care clinics (2 in each arm) and were eligible for but had not yet received the COVID-19 vaccine.
  Percent of participants vaccinated
    number analyzed (Participants) | 659 | 1174 | 1833
    (all) | 31.0 | 34.8 | 33.4

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Vaccination Rate for Eligible Children
Description: Percent of patients who received a COVID-19 vaccine among all children who were eligible for and had not yet been vaccinated for the COVID-19 vaccine during the time of their visit to one of the four participating primary care clinics.
Time Frame: 4 months
Population: The multi-component intervention was introduced in phases at the two intervention clinics to understand the effect of each component of COVID-19 vaccination. Individual participants were counted if they had a clinic visit during a particular phase of the trial at either of the 2 intervention clinics or two standard care clinic. Because of this, the number analyzed for each phase is different from one another and different from the number analyzed.
Measure: Number; unit: Percent of participants vaccinated
Units Other Than Participants: Primary care clinic
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
Number analyzed (Participants) | 2221 | 3529
Number analyzed (Primary care clinic) | 2 | 2
Percent of participants vaccinated
  Phase 1: Community-Tailored Handouts: number analyzed (Participants) | 268 | 406
  Phase 1: Community-Tailored Handouts | 21.3 | 33.5
  Phase 2: Videos Featuring Local Families: number analyzed (Participants) | 281 | 476
  Phase 2: Videos Featuring Local Families | 16.4 | 26.7
  Phase 3: Family-Centered Communication at Primary Care Clinic: number analyzed (Participants) | 442 | 628
  Phase 3: Family-Centered Communication at Primary Care Clinic | 21.9 | 19.4
  Phase 4: Community Health Worker Outreach: number analyzed (Participants) | 1230 | 2019
  Phase 4: Community Health Worker Outreach | 14.4 | 10.6

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Culturally-Tailored COVID-19 Vaccine Uptake Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/2244 | 0/3548
Serious Adverse Events (participants affected / at risk) | 0/2244 | 0/3548
Other Adverse Events (participants affected / at risk) | 0/2244 | 0/3548

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT05293392/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT05293392/ICF_001.pdf